CLINICAL TRIAL: NCT02334878
Title: Autologous Bone Marrow-derived Mesenchymal Stem Cells Versus Tension-free Vaginal Tape for Treatment of Female Stress Urinary Incontinence: An Open-label Clinical Trial
Brief Title: Stem Cell Therapy for Treatment of Female Stress Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Rania Hassan Mostafa, assistant lecturer, Ain Shams Maternity Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU 3098/2014
Record Dates: First submitted 2014-12-21; First posted 2015-01-08 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Urinary Incontinence, Stress
Keywords: Stem Cells; Mesenchymal
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stem cells,Mesenchymal (Experimental): Periurethral injection of autologous bone-marrow derived stem cells.
  Interventions: Biological: Stem Cells,Mesenchymal
- surgery (TVT) (Active Comparator): Tension-free vaginal tape operation: a midurethral sling operation
  Interventions: Procedure: surgery (TVT)

INTERVENTIONS:
Biological: Stem Cells,Mesenchymal — The patient will be placed in lithotomy position. A Foley's catheter (size 18) will be inserted in the urethra, then under local anaesthesia; retrieved cells (total 20- 30 million cells per patient in 10cc syringe) will be injected into the submucosal tissue at the level of the proximal urethra just distal to the bladder neck (guided by stretch on the Foley's catheter), at 3,9,12 o'clock, injecting around 3.5 cc in each site.
  Arms: Stem cells,Mesenchymal
Procedure: surgery (TVT) — A small midurethral incision will be made in the vaginal mucosa, then a polypropylene 40*1cm mesh tape attached to two curved trocars will be passed lateral to the urethra & through the endopelvic fascia into the retropubic space. The trocar will then be passed along the back of the pubic bone, through the rectus fascia, in two small suprapubic skin incisions, then the tension on the tape adjusted & the remaining tape cut off at the level of the skin.
  Arms: surgery (TVT)

SUMMARY:
This study evaluates the effectiveness of mesenchymal stem cells in treatment of stress urinary incontinence due to intrinsic sphincter deficiency; in which the problem is weakness or damage of the sphincter muscle responsible for continence. Mesenchymal stem cells are undifferentiated cells which can undergo self-renewal & differentiation into other cell types like muscle cells; thus can be used to regenerate the damaged sphincter muscles. In this study mesenchymal stem cells will be obtained from bone marrow from the patient, processed, & then re-injected periurethrally. Effectiveness will be compared to that of the surgical treatment (tension-free vaginal tape).

DETAILED DESCRIPTION:
** Study settings : The study is to be held at Ain-Shams University Maternity Hospital - urogynecolgy unit; recruiting the patients from the urogynecology outpatient clinic

** Sample size:

Fifty female patients with stress urinary incontinence due to intrinsic sphincter deficiency will be recruited into two groups; group A including 25 patients will be injected with stem cells, & these will be the patients refusing surgery as a primary line of treatment, or unfit for surgery. Group B; including 25 patients, will undergo the tension-free vaginal tape operation. The sample size is determined according to the following equation:

[ P1( 100-P1) + P2( 100-P2) ] / (P2 - P1)2 where; Power of the test = 80% Confidence level = 95% Alpha error = 5% Assuming success rate for the preferably used intervention "tension-free vaginal tape" in patients with intrinsic sphincter deficiency P1=80% ( Schierlitz et al, 2008).

Assuming success rate for stem cell therapy P2= 90% ( Smaldone et al, 2009).

** Intervention:

1. Consent Informed consent will be taken according to World Medical Association (WMA) Declaration of Helsinki; the Ethical Principles for Medical Research Involving Human Subjects.
2. History Full medical history will be taken from each patient, together with detailed history as regards voiding habits, incontinence, voiding dysfunction, urinary infection. Questionnaire about incontinence, & questionnaire about quality of life will be obtained.
3. Examination Complete physical and pelvic examination to evaluate the presence of stress urinary incontinence, & to exclude patients with marked hypermobility of the urethra, or severe cystocele or rectocele.
4. Urodynamic study A multi-channel urodynamic study using Euet Sensik ® will be performed including cystometry, urethral pressure measurement, abdominal leak point pressure (ALPP) measurement, & residual urine measurement. Patients with stress urinary incontinence due to intrinsic sphincter deficiency will be selected. Criteria for selection are: absence of involuntary contractions during leakage caused by a stress maneuver; low ALPP (<60 cmH2O); & maximum urethral closure pressure (MUCP) <20-30 cmH2O. Patients with voiding dysfunction will be excluded (residual urine volume >100ml).
5. Cells retrieval, culture, & processing:

   * Bone marrow aspiration:

   -Site: posterior superior iliac crest.

   -Procedure: The patient is placed in the lateral decubitus position, with the top leg flexed and the lower leg straight. The iliac crest is palpated, and the preferred sampling site is marked with a pen. Aseptic technique is employed, including sterile gloves and gown. The site is prepared with an antiseptic (povidone-iodine), scrubbed, and draped, exposing only the site to be sampled. The skin and the underlying tissue to the periosteum are infiltrated with a local anaesthetic (approximately 10 mL of 1% Xylocaine [lidocaine]). A 10-mL syringe with a 25-gauge needle is used to inject an initial 0.5 mL directly under the skin, raising a wheal. A 22-gauge needle is used to penetrate deeper into the subcutaneous tissue and the underlying periosteum, an area roughly 1 cm in diameter. A skin incision is made with a small surgical blade, through which the bone marrow aspiration needle, with a stylet locked in place, is inserted. Once the needle contacts the bone, it is advanced by slowly rotating clockwise and counter clockwise until the cortical bone is penetrated and the marrow cavity is entered. The depth of the penetration should not extend beyond an initial 1cm. Once within the marrow cavity, the stylet is removed. Using a 20 mL syringe, approximately 5 mL of bone marrow are aspirated. Subsequent specimens are obtained by attaching a separate syringe, collecting 5 mL at a time. The samples are then transferred into an ethylenediaminetetraacetic acid (EDTA) -containing tube. The marrow needle is removed, and pressure is applied to the aspiration site with gauze until any bleeding stops.

   * Cells processing & culture:

   - Mononuclear cells (MNCs) will be isolated by density gradient centrifugation using Ficol/Hypaque.

   - Mesenchymal stem cells (MSCs) will be isolated through plastic adherence by the seeding of MNCs in T25 tissue culture flasks in complete culture media (DMEM, 1% antibiotics/antifungal, 20% autologous serum). Flasks will be incubated at 37ºC in CO2 incubator for 3-5 days.

   - After 5 days, flasks will be evaluated under inverted microscope for the number and morphology of MSCs. Non-adherent cells will be discarded and medium replenished.

   - Half of the medium will be changed every 3 days.

   - Flasks will be evaluated until cells reach about 80-90% confluence.
   * MSCs will be harvested using Trypsin-EDTA (0.25%) for 5 minutes. Afterwards, trypsin action will be stopped by the addition of autologous serum.
   * MSCs will be washed using phosphate buffered saline (PBS), counted, tested for viability using trypan blue exclusion test.
   * MSC will be identified using immunophenotypic markers (positive for CD44 and negative for CD34).
   * Cells will be suspended in sterile saline, a minimum of 20 X 106 MSCs cells in a 10 cc syringe, ready for injection.

   Quality control check for the sterility by the performance of bacterial aerobic and anaerobic cultures will be done to ensure the complete aseptic conditions during the specimen retrieval, preparation, storage, and injection. (Gunetti et al., 2012)
6. Injection of cells:

   The patient will be placed in lithotomy position. A Foley's catheter (size 18) will be inserted in the urethra, then under local anaesthesia; retrieved cells (total 20- 30 million cells per patient in 10cc syringe) (Sebe et al., 2011) will be injected into the submucosal tissue at the level of the proximal urethra just distal to the bladder neck (guided by stretch on the Foley's catheter), at 3,9,12 o'clock, injecting around 3.5 cc in each site.
7. Tension-free vaginal tape (TVT):

   Another 25 patients will undergo surgical intervention, which is the "tension-free vaginal tape" operation at the obstetrics & gynecology department - Ain Shams Maternity Hospital - urogynecology unit. In this technique, a small midurethral incision will be made in the vaginal mucosa, then a polypropylene 40*1cm mesh tape attached to two curved trocars will be passed lateral to the urethra & through the endopelvic fascia into the retropubic space. The trocar will then be passed along the back of the pubic bone, through the rectus fascia, in two small suprapubic skin incisions, then the tension on the tape adjusted & the remaining tape cut off at the level of the skin.
8. Follow up:

Follow up visits will be conducted at 3months, 6months, 9months, and 12months after therapy. Clinical examination, incontinence questionnaire, quality of life questionnaire, & urodynamic study will be done.

** Data collection & recording:

Each patient will have a case record form (CRF) in which the following data will be recorded:

* Age, parity
* Body mass index (BMI).
* Type of intervention (stem cell therapy or TVT)
* International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) on admission & 3m, 6m, 9m, 12m post-injection.
* Incontinence Quality of Life (I-QOL) Instrument Score on admission & 3m, 6m, 9m, 12m post-injection.
* Cough test on admission & 3m, 6m, 9m, 12m post-injection.
* Urodynamic study on admission & 3m, 6m, 9m, 12m post-injection.

  * Statistical analysis:

Descriptive statistics for measured variables will be expressed as range, mean and standard deviation (for metric data); range, median and interquartile range (for discrete data); and number and proportions (for categorical data). Pre-injection & post-injection findings will be compared using the t-test or the Wilcoxon test depending on whether the measured parameters were Gaussian variables. A P-value of 0.05 or less will be considered statistically significant.

** Ethical considerations:

1. Delegation of investigator responsibilities:

   The investigator will ensure that all persons assisting with the trial are adequately informed about the protocol, & their trial-related duties and functions. The investigator will maintain a list of sub-investigators and other appropriately qualified person to whom he or she has delegated significant trial-related duties.
2. Patient information and informed consent Before being admitted to the clinical study, the patient must consent to participate after the nature, scope, and possible consequences of the clinical study have been explained in a form understandable to her. An informed consent document, in Arabic language, contains all locally required elements and specifies who informed the patient. After reading the informed consent document, the patient must give consent in writing. The patient's consent must be confirmed at the time of consent by the personally dated signature of the patient and by the personally dated signature of the person conducting the informed consent discussions. If the patient is unable to read, oral presentation and explanation of the written informed consent form and information to be supplied to patients must take place in the presence of an impartial witness. Consent must be confirmed at the time of consent orally and by the personally dated signature of the patient or by a local legally recognized alternative (e.g., the patient's thumbprint or mark). The witness and the person conducting the informed consent discussions must also sign and personally date the consent document. The original signed consent document will be retained by the investigator. The investigator will not undertake any measures specifically required only for the clinical study until valid consent has been obtained.
3. Confidentiality Only the patient number and patient initials will be recorded in the CRF, and if the patients name appears on any other document, it must be kept in privacy by the investigators. The investigator will maintain a personal patient identification list (patient numbers with the corresponding patient names) to enable records to be identified.
4. Protocol approval Before the beginning of the study and in accordance with the local regulation followed, the protocol and all corresponding documents will be declared for ethical and research approval by the council of ob/gyn department, Ain Shams University; according to the WMA Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of stress urinary incontinence
* Urodynamic study showing stress urinary incontinence due to intrinsic sphincter deficiency

Exclusion Criteria:

* Pregnant females
* Hypermobility of the urethra
* Mild cases (treatment is mainly physiotherapy & pelvic floor exercises)
* Urge incontinence / Urodynamic study showing detrusor instability
* Current urinary infection
* Current severe cystocele or rectocele
* History of previous synthetic, biologic or fascial sub-urethral sling or any other surgery on external genitalia, bladder neck, bladder or urethra
* Voiding dysfunction (post-void residual volume >100cc)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
change in cough test & urodynamic study as a measure of efficacy of treatment | before & after therapy each 3 months for one year (at 3m, 6m, 9m, 12m post-injection).
  cough test: as positive or negative leakage with cough. Urodynamic study: changes in abdominal leak point pressure, and changes in maximum urethral closure pressure

SECONDARY OUTCOMES:
Quality of life as measured by the Incontinence Quality of Life (I-QOL) Instrument Score | before & after therapy each 3 months for one year (at 3m, 6m, 9m, 12m post-injection).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A El-Nazer, PhD, Study Chair — Ain Shams University Maternity Hospital; Abdel-Latif G El-Kholy, PhD, Study Director — Ain Shams University Maternity Hospital; Mostafa F Gomaa, PhD, Study Director — Ain Shams University Maternity Hospital
Locations (1):
- Maternity hospital, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No